CLINICAL TRIAL: NCT05192369
Title: A Four-Arm, Randomized, Crossover, Placebo and Active Controlled Study for the Evaluation of the Effect of Therapeutic and Supratherapeutic Doses of CTP-543 on the QT/QTc Intervals in Healthy Volunteers
Brief Title: A Randomized Study to Evaluate the Effects of CTP-543 on the QT/QTc Intervals in Health Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CP543.1010
Record Dates: First submitted 2022-01-05; First posted 2022-01-14 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Healthy Volunteers
Keywords: CTP-543
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A: Therapeutic Dose (Experimental): Single oral dose of 12mg CTP-543
  Interventions: Drug: CTP-543
- Treatment B: Supratherapeutic Dose (Experimental): Single oral dose of 48mg CTP-543
  Interventions: Drug: CTP-543
- Treatment D: Placebo (Placebo Comparator): Single oral dose of 1 Placebo tablet
  Interventions: Drug: Placebo
- Treatment C: Positive Control (Active Comparator): Single oral dose of 400mg Moxifloxacin
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: CTP-543 — CTP-543 12 mg (1 x 12 mg tablet), dosed with water
  Arms: Treatment A: Therapeutic Dose
Drug: CTP-543 — CTP-543 48 mg (4 x 12 mg tablet) dosed with water
  Arms: Treatment B: Supratherapeutic Dose
Drug: Moxifloxacin — Moxifloxacin (1 x 400 mg tablet) dosed with water
  Arms: Treatment C: Positive Control
Drug: Placebo — Placebo (1 tablet) dosed with water
  Arms: Treatment D: Placebo

SUMMARY:
This is a four-arm, randomized, crossover, placebo and active controlled study to evaluate of the effect of therapeutic and supratherapeutic doses of CTP-543 on the QT/QTc intervals in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking, adult males or females aged 18-60
* Body mass index of 18 to 32 mg/m2 at Screening
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or Electrocardiograms (ECGs)
* If of reproductive age, willing and able to use a medically highly effective form of birth control 30 days prior to first dose, during the study and for 30 days following last dose of study medication
* Understands the study procedures in the informed consent form and be willing and able to comply with the protocol

Exclusion Criteria:

* History or presence of clinically significant medical or psychiatric condition or disease
* History of any illness that might confound the results of the study or poses an additional risk to the subject by their participation in the study
* History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing
* History of prolonged QT syndrome or a Corrected QT-interval (QTc) with Fridericia's correction (QTcF) > 450 msec for males or QTcF > 470 msec for females obtained at Screening visit or prior to the first dosing
* Females who are nursing, pregnant, or planning to become pregnant while in the study, and for 30 days after last dose of study drug
* Positive results at Screening for human immunodeficiency virus, hepatitis B surface antigen or hepatitis C virus
* A positive test or history of incompletely treated or untreated tuberculosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
TQT Analysis | Before dosing (pre-dose) through 24 hours post-dose on Day 1, Day 4, Day 7, and Day 10
  Analysis of the change from pre-dose-averaged baseline Fridericia's corrected QT interval (QTcF) at each post-dose timepoint

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology of Miami, LLC, Miami, Florida, United States